CLINICAL TRIAL: NCT02970097
Title: Comparison Between Infraclavicular Brachial Plexus Block Versus Local Infiltration for Postoperative Analgesia After Wrist Arthroscopy, a Prospective Randomized Open Label Study
Brief Title: Single Shot Infraclavicular Brachial Plexus Block vs Local Infiltration After Wrist Arthroscopy Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 825465
Record Dates: First submitted 2016-10-24; First posted 2016-11-21 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Wrist Injuries; Postoperative Pain Control
Keywords: infraclavicular brachial plexus block; wrist arthroscopy; quality of recovery score; pain score; modified sleep quality assessment
MeSH Terms: conditions — Wrist Injuries | interventions — Ropivacaine; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single shot IBP block (Active Comparator): Subjects will receive single shot infraclavicular brachial plexus block with 20ml bolus of 0.5% ropivicaine given preoperatively to help with operative and postoperative pain
  Interventions: Drug: 20ml bolus of 0.5% ropivicaine; Drug: Midazolam; Drug: Fentanyl
- local infiltration (Active Comparator): Subjects will receive local infiltration into portal space and joint space with 10ml of 0.5% ropivicaine given intraoperatively to help with operative and postoperative pain
  Interventions: Drug: 10 ml of 0.5% ropivicaine

INTERVENTIONS:
Drug: 20ml bolus of 0.5% ropivicaine — local anesthetic
  Other Names: Naropin
  Arms: single shot IBP block
Drug: 10 ml of 0.5% ropivicaine — local anesthetic
  Other Names: Naropin
  Arms: local infiltration
Drug: Midazolam — 1-2 mg of medication given intravenously before nerve block
  Other Names: Versed
  Arms: single shot IBP block
Drug: Fentanyl — 50-100 mcg of medication given intravenously before nerve block
  Other Names: Sublimaze; Actiq; Durogesic; Fentora
  Arms: single shot IBP block

SUMMARY:
The purpose of this study is to compare infraclavicular brachial plexus shot single shot block to local infiltration done in adult patients having wrist arthroscopy surgery. Visual analogue scores, opioid consumption, quality of recovery and quality of sleep up to 72 hours post operatively will be used for comparison.

DETAILED DESCRIPTION:
If the patient is willing to participate and signs the consent, he/she will be randomized to one of the two treatment groups:

1. Single shot block
2. Local Infiltration

In the institution investigators usually advocate for regional anesthesia and intravenous sedation for the repair of open fracture of the distal radius.

Patients will be monitored during block performance with standard ASA monitors. All patients will receive 2 L of oxygen via a nasal cannula. Sedatives will be titrated to effect. Midazolam 1-2 mg, and fentanyl 50-100 mcg will be used for sedation.

Block time out will be preformed according to standard operating procedure. All blocks will be done under ultrasound guidance. Sonosite S nerve machine will be used with a low frequency curvilinear (C5) US probe with 2-5 MHZ frequency. Both single shot and local infiltration will be performed according to the SOP in the department. Ultrasound survey of the deltopectoral groove below the clavicle will take place. The axillary artery and the three cords (posterior, medial and lateral) of the brachial plexus will be identified in short axis view deeper to the pectoralis minor muscle.

For single shot blocks: A 4 inch 21 gauge single shot (B-Braun) needle will be introduced in-plane towards the posterior cord of the brachial plexus and 1-2 mL of dextrose 5% (D5%) bolus will be used to verify correct placement of the needle in the vicinity of the posterior cord and adequate spread pattern to both lateral and medical cord. 20 ml of of Ropivicaine 0.5% will be injected through the needle with intermittent aspiration after each 5 ml bolus injection.

For local infiltration: At the end of surgery, surgeon will inject 10 ml of Ropivacaine 0.5% into the arthroscopy portals and the wrist. Specifically, 1 ml to 2 ml of Ropivacaine 0.5% will be injected into each portal with the remainder of the volume injected into the joint space itself.

Block success will be defined as a change in cutaneous sensation to touch with an alcohol pad in the posterior, medial and lateral cord distribution over the forearm and the hand within 30min after injection. Subjects with successful catheter placement per protocol and nerve block onset will be retained in the study. Subjects with a failed catheter insertion or misplaced catheter indicated by a lack of sensory changes will have their catheter replaced or will be single shot blocked and withdrawn from the study.

Intraoperative sedation will consist of intermittent boluses of midazolam (1-2 mg), fentanyl (50-100 mcg) and propofol infusion, titrates to sedation and patient comfort (25-50 mcg/kg/min).

All patients will receive prophylaxis for postoperative nausea and vomiting (PONV) during surgery. The protocol for prophylaxis against PONV includes administration of 4 mg of dexamethasone after induction of anesthesia and 4 mg of ondansetron 20 minutes before recovery from anesthesia. Dexamethasone is withheld if the patient has poorly controlled diabetes mellitus (DM). Uncontrolled DM will be defined as random blood glucose above 250 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for wrist arthroscopy
* American Society of Anesthesiologists (ASA) physical status I -III
* Mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Patient younger than 18 years old
* Allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone and any of the drugs included in the standard of care
* Patients opting to go under light anesthesia and those refusing the block
* Chronic pain syndromes; Patients will be defined to have chronic pain if they are using regular daily doses of systemic narcotics for the past 6 months prior to the surgery
* BMI of 40 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Pain Scores as measured by the Visual Analog Scale | 72 hours
  Pain scores at rest and with movement.
Participants need for pain relief as measured by opiate consumption | 72 hours
  Amount of opiate consumption

SECONDARY OUTCOMES:
Quality of recovery score | 7 days
  Score of QoR survey to determine recovery status
quality of sleep as measured by modified Pittsburgh Sleep Quality Index | 72 hours
  a 9-question survey in which patients report how often sleep-related problems occur on a scale of 0 to 3
Range of motion as measured by the Disability assessment of shoulder and hand questionnaire | 3 months
  Dash questionnaire to measure range of motion of the wrist and fingers 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Elkassabany, MD, Principal Investigator — University of Pennsylvania, Anesthesia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States